CLINICAL TRIAL: NCT00645541
Title: Axillary Reverse Mapping for Invasive Carcinoma of the Breast
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2007-0951
Record Dates: First submitted 2008-03-25; First posted 2008-03-27 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-08

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Carcinoma of the Breast; Lymph Nodes; Lymphazurin; Axillary Reverse Mapping
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Axillary Reverse Mapping (ARM) (Experimental)
  Interventions: Procedure: Axillary Reverse Mapping

INTERVENTIONS:
Procedure: Axillary Reverse Mapping — Lymphazurin, isosulfan blue dye, injected into arm then a standard axillary lymph node surgery to remove any blue dyed lymph nodes found (lymph nodes that have traveled down the drainage pathways).

SUMMARY:
Primary Objectives:

* To determine the feasibility of axillary reverse mapping (ARM) in patients undergoing axillary lymph node dissection for breast cancer therapy.
* To determine the incidence of breast cancer metastasis in lymph nodes draining in the arm as identified by axillary reverse mapping.
* To determine the safety of axillary reverse mapping.

DETAILED DESCRIPTION:
Lymphazurin is a blue dye used usually in breast cancer surgery to trace the drainage pathway that flows to lymph nodes. The dye will travel to the lymph system and will end up in the lymph nodes that are draining the arm.

In this study, lymphazurin will be used to find the drainage routes from your arm, rather than your breast.

AXILLARY REVERSE MAPPING:

Before axillary lymph node surgery, your surgeon will inject lymphazurin into your arm. Your surgeon will watch how the dye flows and find the channels and nodes draining the arm. You will then have standard axillary lymph node (lymph nodes found under the arm) surgery. Any lymph nodes found that are dyed blue (lymph nodes that have traveled down the drainage pathways) that would normally be removed will be removed and sent to the pathology department. Pathologists will check the nodes to see if they have breast cancer cells in them. Also as part of routine care, all other axillary lymph nodes draining the breast will be removed and checked for breast cancer cells.

This is an investigational study. Lymphazurin is FDA approved and commercially available. The use of lymphazurin with axillary reverse mapping is investigational.

Up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive carcinoma of the breast planning to undergo axillary lymph node dissection at M. D. Anderson Cancer Center.
* Eastern Cooperative Oncology Group (ECOG) performance status of equal to or less than 3.

Exclusion Criteria:

* Patients with known allergies to blue dye or other contraindications to Lymphazurin.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2008-03; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
Identification Rate for Feasibility of ARM in Patients Undergoing Axillary Lymph Node Dissection for breast cancer therapy | 2 years for overall study
  Axillary reverse mapping (ARM) performed using 2 - 5cc of isosulfan blue, injected into the inner arm prior to skin incision for the axillary lymph node dissection. Blue channels identified during surgery and locations compared to axillary vein. Any blue nodes within the standard axillary lymph node dissection field removed then sent to pathology as a separate specimen labeled "axillary reverse mapping nodes" and evaluated with serial sectioning, and hematoxylin-eosin stain (H&E) as well as immunohistochemistry.

SECONDARY OUTCOMES:
Incidence of breast cancer metastasis in lymph nodes draining in the arm as identified by ARM | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Funda Meric-Bernstam, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org